CLINICAL TRIAL: NCT05707195
Title: Improvement the Quality of Care Through the Implementation of a Learning From Excellence Program in a Pediatric Intensive Care Unit
Brief Title: Learning Excellence Program and Improvement of Quality Care
Acronym: RECOMPENSE
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0020
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-02

CONDITIONS: Satisfaction, Patient
MeSH Terms: conditions — Patient Satisfaction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental:children hospitalized in pediatric intensive care unit: All parents of children aged 0 to 18 who have been hospitalized in the pediatric intensive care unit over a period of 24 months will be offered the study.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A questionnaire is offered to parents of patients who meet the eligibility criteria and who have given their non-objection.
  This questionnaire aims to evaluate the quality of care perceived by the parents of children hospitalized in the pediatric intensive care unit

SUMMARY:
Improving the quality of care is a daily goal in pediatric intensive care units. Measuring patient and family satisfaction is recognized as an indicator of quality of care. A validated questionnaire was specially developed to study parental satisfaction in pediatric intensive care units. A positive multi-professional analysis of clinical situations, using appreciative inquiry, within a health service can create new opportunities for learning and innovation. The establishment of such a Learning From Excellence (LfE) program tends to increase the well-being and self-confidence of caregivers and promotes dynamic learning educational programs, including simulation.

It therefore seems important to assess the improvement in the quality of care in pediatric intensive care following the implementation of a Learning From Excellence program allowing positive reflection on practices as well as innovations within the service.

ELIGIBILITY:
Inclusion Criteria:

* All parents of children aged 0 to 18 who have been hospitalized in the pediatric intensive care unit over a period of 24 months once the research has been authorized and started

Exclusion Criteria:

* Parents unable to answer the questionnaire because they do not speak French
* Parents of children who died during their stay in the pediatric intensive care unit

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Parents of children aged 0 to 18 who have been hospitalized in the pediatric intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the quality of care. | Day 1, the day of discharge from hospital
  Satisfaction will be measured via the EMpowerment of Parents in THe Intensive Care questionnaire score (EMPATHIC-65 questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Breinig, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No